CLINICAL TRIAL: NCT06312722
Title: Safety and Effectiveness of the Optilume® BPH Catheter System in a Post-Market Study
Acronym: PEAK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Urotronic Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PR1309
Record Dates: First submitted 2024-03-08; First posted 2024-03-15 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Benign Prostatic Hyperplasia
MeSH Terms: conditions — Prostatic Hyperplasia

STUDY DESIGN:
Intervention Model Description: Prospective, single-arm, multi-center, post market clinical trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Study Arm (Other): Optilume BPH Catheter System
  Interventions: Device: Optilume® BPH Catheter System

INTERVENTIONS:
Device: Optilume® BPH Catheter System — The Optilume BPH Catheter System is a combination drug/device minimally invasive surgical therapy (MIST) comprised of an uncoated pre-dilation balloon catheter and a separate drug coated balloon (DCB) catheter. The distal end of each catheter has a semi-compliant, inflatable, double lobe balloon that is used to dilate the prostate. The double-lobe DCB catheter is coated with a proprietary coating containing the active pharmaceutical agent paclitaxel. The drug coating covers the working length of the balloon body.

SUMMARY:
The goal of this clinical trial is to verify the continued safety and effectiveness for the Optilume BPH Catheter System.

DETAILED DESCRIPTION:
The goal of this clinical trial is to verify the continued safety and effectiveness for the Optilume BPH Catheter System.

STUDY ENDPOINTS

Primary Efficacy Endpoint:

The primary efficacy endpoint is the average IPSS improvement from baseline to 12 months.

Primary Safety Endpoint:

The primary safety endpoint is the freedom from composite treatment-related adverse SAEs.

Key Secondary Safety Endpoint (Semen Sub-Study Only):

The average change from baseline in sperm concentration at 13 weeks (3 months) post-procedure will be compared against a performance goal of -30% (30% decrease from baseline).

Ancillary Endpoints:

Ancillary Safety Endpoint:

1. Frequency and severity of treatment-related AEs Adverse events will be collected and assessed for relatedness to the device and the procedure as well as for severity. The Clavien-Dindo severity grading scale is a commonly used criteria in the urology community. An independent medical monitor will adjudicate all treatment-related events.
2. Frequency and severity of all AEs All adverse events will be summarized and reported, regardless of relatedness to the device or procedure.
3. Change from baseline in semen characteristics over time (semen sub-study only) Semen characteristics (concentration, count, motility) will be summarized at each follow-up, including change from baseline values. Reported values for each subject will represent an average of 2 samples collected at each timepoint. Summary statistics will be based on reported values for each subject at each timepoint.
4. Proportion of subjects experiencing ≥50% decrease in sperm concentration from baseline The proportion of subjects experiencing ≥50% decrease in sperm concentration from baseline to 3, 6 and 12 months will be reported.

   Ancillary Efficacy Endpoints:
5. Improvement in IPSS over time The IPSS tool is the most commonly reported symptom score for obstructive urinary symptoms secondary to BPH. Average IPSS scores, absolute change from baseline, and percent change from baseline will be reported at each follow-up timepoint.
6. Improvement in ICS male SF over time The International Continence Society (ICS) male short form (SF) has three domains to assess urinary symptoms; voiding symptoms (e.g., hesitancy, incomplete voiding, etc.), storage symptoms (e.g., frequency), and leakage symptoms. Average total scores and average scores for each domain, along with changes from baseline, will be reported at each follow-up timepoint.
7. Improvement in Qmax over time Uroflowmetry represents an objective measure of relief of obstruction. Average peak urinary flow rate (Qmax) and change from baseline will be reported at each follow-up timepoint.
8. Improvement in PVR over time Residual urine in the bladder due to incomplete emptying is an important clinical consideration in subjects with obstructive BPH. Average PVR and change from baseline will be reported at each follow-up timepoint.
9. Freedom from repeat intervention (time-to-event) The proportion of subjects free from repeat surgical or endoscopic intervention for BPH will be reported over time utilizing the Kaplan-Meier method.

ELIGIBILITY:
Inclusion Criteria:

1. Male subject ≥ 50 years old
2. Diagnosed with lower urinary tract symptoms (LUTS) secondary to obstructive benign prostatic hyperplasia (BPH)
3. Able to be treated with the Optilume BPH Catheter System in accordance with the Instructions for Use
4. Prostate volume < 80 g with a prostatic urethral length between 32-55 mm as determined by trans-rectal ultrasound (TRUS)
5. International Prostate Symptom Score (IPSS) ≥ 13
6. Peak urinary flow rate (Qmax) 5-15 mL/sec with minimum voided volume of 125 mL
7. Willing to provide informed consent and comply with protocol required follow-up

Exclusion Criteria:

1. Unwilling to abstain from sexual intercourse or use a condom for 30 days post-procedure and utilize a highly effective contraceptive for at least 12 months post-procedure
2. Presence of an artificial urinary sphincter, penile prosthesis, or stent(s) in the urethra or prostate
3. Any prior minimally invasive intervention (e.g., TUNA, Balloon, Microwave, Rezūm, UroLift) or surgical intervention of the prostate
4. Confirmed or suspected malignancy of prostate or bladder. Negative prostate biopsy required within 6 months of enrollment if PSA at baseline is > 4 ng/mL with free PSA < 25%.
5. Active urinary tract infection (UTI) confirmed by culture
6. Neurogenic bladder or sphincter abnormalities or neurological disorders that might affect bladder or sphincter function
7. History of overt urinary incontinence requiring the use of pads
8. Previous or current diagnosis of urethral strictures, bladder neck contracture or detrusor muscle spasms
9. Current post-void residual volume (PVR) > 300 mL or catheter dependent bladder drainage
10. Known poor detrusor muscle function (e.g., Qmax < 5 mL/sec)
11. Active bladder, ureteral, or urethral stones or stone passage within the last 3 months
12. Current poorly controlled diabetes (i.e., hemoglobin A1c ≥ 8%)
13. Anatomy (e.g., presence of false passage or size of meatus) is not suitable for treatment with the Optilume BPH Catheter System
14. Obstructive median lobe in the opinion of the investigator

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — BPH is a disease of the prostate
Enrollment: 92 (Estimated)
Dates: Start 2024-02-07 (Actual); Primary Completion 2031-02-07 (Estimated); Study Completion 2031-02-07 (Estimated)

PRIMARY OUTCOMES:
Change in International Prostate Symptom Score (IPSS) | Baseline to 12 months
  The primary efficacy endpoint is the average IPSS improvement from baseline to 12 months.
  The first seven questions in the International Prostate Symptom Score (IPSS) questionnaire address frequency, nocturia, weak urinary stream, hesitancy, intermittence, incomplete emptying, and urgency, and scored on a 6-point scale (0 to 5). The IPSS can be interpreted as follows: 0-7 mildly symptomatic, 8-19 moderately symptomatic, and 20-35 severely symptomatic.
Rate of a composite of treatment-related serious adverse events (SAEs) | 3 months
  The primary safety endpoint is the rate of a composite of the specified treatment-related serious adverse events through 3 months post-treatment:
  * De novo severe urinary retention lasting >14 days post-procedure
  * De novo severe stress urinary incontinence requiring surgical management
  * Formation of a fistula between the rectum and urethra
  * Perforation of the rectum or GI tract
  * Bleeding requiring transfusion or endoscopic intervention

SECONDARY OUTCOMES:
Change in Sperm Concentration | Baseline to 3 months
  For the Semen Sub-Study, the average change from baseline in sperm concentration at 13 weeks (3 months) post-procedure will be compared against a performance goal of -30% (30% decrease from baseline).

CONTACTS AND LOCATIONS:
Overall Officials: Steven Kaplan, MD, FACS, Principal Investigator — Professor of Urology
Locations (5):
- United States (5):
  - Arkansas Urology, Little Rock, Arkansas
  - Florida Urology Partners, LLP, Tampa, Florida
  - Ochsner LSU Health Shreveport - Regional Urology, Shreveport, Louisiana
  - Sheldon Freedman MD, Ltd, Las Vegas, Nevada
  - Midtown Urology Associates, Austin, Texas

IPD SHARING:
Plan to Share IPD: No